CLINICAL TRIAL: NCT02910115
Title: Can Cooling the Uterus During Cesarean Delivery Reduce Blood Loss, Reduce Drug Use, and Decrease the Risk for Hysterectomy in Women With Dysfunctional Labor?
Brief Title: Cooling the Uterus in C-section After Dysfunctional Labor
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in acquiring patients in a reasonable amount of time.
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: 015-028
Record Dates: First submitted 2016-01-14; First posted 2016-09-21 (Estimated); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Blood Loss; Dysfunctional Labor; Uterine Atony
MeSH Terms: conditions — Hemorrhage; Dystocia; Uterine Inertia | interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Other): Following delivery of the fetus patients in the control group will have Pitocin® administered to them intravenously according to the usual protocol. The uterus may be wrapped lap sponges soaked in room-temperature saline while the uterine incision is closed per the attending obstetrician's usual practice. At the discretion of the attending obstetrician additional uterotonic medications (Pitocin®, Methergine® Cytotec® and/or Hemabate®) may be given to improve uterine contraction.
  Interventions: Drug: Pitocin
- Study Group (Experimental): Following delivery of the fetus, patients in the study group also will have Pitocin® administered to them according to the usual protocol.
  Immediately following delivery of the fetus the uterus will be externalized in the usual fashion and the body of the uterus cephalad to the hysterotomy incision will be wrapped in cold laparotomy sponges saturated in sterile, iced normal saline. The skin of the abdomen will be draped to prevent contact with the cold towels. Additional uterotonic medications may be given at the discretion of the attending obstetrician.
  Interventions: Other: Cold laparotomy sponges; Drug: Pitocin

INTERVENTIONS:
Other: Cold laparotomy sponges — Cold laparotomy sponges are lap sponges that are saturated in sterile, iced normal saline
  Other Names: cold lap sponges
  Arms: Study Group
Drug: Pitocin — Pitocin is administered intravenously according to the usual protocol.
  Other Names: IV Oxytocin

SUMMARY:
The objective of the study is to demonstrate whether cooling the uterine smooth muscle during cesarean section (following delivery of the fetus) will promote better uterine contraction and involution resulting in lower blood loss, use of fewer uterotonic medications, and fewer hysterectomies following cesarean section for dysfunctional labor.

DETAILED DESCRIPTION:
Two hundred patients will be drawn from all pregnant women who require a cesarean delivery for dysfunctional labor. Dysfunctional labor will be defined as cervical dilation of 3 or more centimeters, in active labor without cervical change for 2 or more hours. Patients will be randomly assigned to the study group or the control group, and each group will have 100 patients.

Following the delivery of the fetus, patients in the control group will have IV Pitocin administered per the usual protocol and the uterus will be wrapped in lab sponges soaked in room-temperature saline while the uterine incision is closed per the attending obstetrician's usual practice. Additional utero-tonic medications may be given to improve uterine contraction.

In the study group, following the delivery of the fetus, the uterus will be externalized in the usual fashion, except the uterus will be wrapped with lap sponges saturated in sterile, iced normal saline. Additional utero-tonic medications may also be given in the study group to improve uterine contraction.

Immediately after the delivery of the fetus and prior to the delivery of the placenta, the amniotic fluid and blood on the surgical field will be aspirated into the suction canister. This amount of fluid in the suction canister will be noted and subtracted from the amount of fluid in the canister at the conclusion of the surgery.

At the conclusion of the surgery, blood loss will be calculated by measuring the content of blood in the suction canister, and by weighing the surgical sponges. Post surgical vaginal bleeding will be monitored and calculated until the patient is discharged from the labor and delivery unit. Use of utero-tonic medications will be recorded.

At the conclusion of the study, the amount of blood loss and utero-tonic drugs between the control and study groups will be compared. The need for additional surgeries, such as a hysterectomy or D&C, will be compared between the two groups.

ELIGIBILITY:
Inclusion criteria:

* pregnant women of any age
* gravidity and gestational duration who present for cesarean section and who have given informed consent to be in the study.

Exclusion criteria:

* Women who refuse to be in the study
* women who are unable to consent due to emergent nature of the cesarean section
* women who are unable to understand the nature of the study due to mental illness, mental retardation, medical condition, or other communication barrier will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-05-14 (Actual); Primary Completion 2017-11-10 (Actual); Study Completion 2018-11-10 (Actual)

PRIMARY OUTCOMES:
Estimated Blood Loss | up to 24 hours after surgery

SECONDARY OUTCOMES:
Change in Hematocrit | up to 24 hours after surgery
Need for use of uterotonic medications | during cesarean section

CONTACTS AND LOCATIONS:
Overall Officials: Jack Stecher, MD, Principal Investigator — BUMC Labor and Delivery

IPD SHARING:
Plan to Share IPD: No